CLINICAL TRIAL: NCT06358313
Title: Concomitant Use of Clopidogrel With Atorvastatin or Rosuvastatin in Patients With Moderate and Moderate-to-severe Stroke, a Randomized Controlled Single-blinded Trial
Brief Title: Concomitant Use of Clopidogrel With Atorvastatin or Rosuvastatin in Patients With Moderate and Moderate-to-severe Stroke
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Kafrelsheikh University (Other)
Responsible Party: Principal Investigator, Mohamed G. zeinhom, MD, principal investigator, Kafrelsheikh University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 0023098816
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Ischemic Stroke
Keywords: atorvastatin; rosuvastatin; clopidogrel; stroke; Egypt
MeSH Terms: conditions — Ischemic Stroke; Stroke | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Intervention Model Description: The study will be composed of 2 arms atorvastatin arm, which consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and the rosuvastatin arm consisted of 300 patients who received 20 mg rosuvastatin daily for 3 months, All the patients in the two groups received an open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Our study was single-blinded to the investigators; an independent statistician generated a computer-generated randomization chart with a block size of four in a one-to-one ratio, and participants were randomly assigned to receive either atorvastatin or rosuvastatin by a specially trained and qualified nurse. None of the investigators included in the study knew the patients' assignments. We prepared Sequentially numbered opaque sealed envelopes and 600 labels for each drug labeled Drug A or B. According to the randomization chart, put them into envelopes numbered 1 to 600. Envelopes were attached to the patient's files. Patients were given enrollment numbers starting from 1, which were mentioned in their files. Files with the same number as the patient enrolment number were opened and the patients were assigned to receive drugs A or B. Drug A included atorvastatin bills, and Drug B included rosuvastatin bills. The statistical analysis was performed by an independent statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- atorvastatin (Active Comparator): The Atorvastatin arm consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, an open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months
  Interventions: Drug: Atorvastatin 40mg
- rosuvastatin (Active Comparator): The rosuvastatin arm consisted of 300 patients who received 20 mg daily rosuvastatin for 3 months and an open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months
  Interventions: Drug: Rosuvastatin 20mg

INTERVENTIONS:
Drug: Atorvastatin 40mg — The atorvastatin group consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Other Names: group A
  Arms: atorvastatin
Drug: Rosuvastatin 20mg — The rosuvastatin group consisted of 300 patients who received 40 mg daily rosuvastatin for 3 months, and open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.
  Other Names: group B
  Arms: rosuvastatin

SUMMARY:
Along with the current clinical trial, the impact of adding atorvastatin or rosuvastatin in the first 24 hours on the clinical outcomes of first-ever moderate and moderate to severe stroke patients treated with clopidogrel and aspirin assessed through NIHSS, mRS, and possible adverse effects.

DETAILED DESCRIPTION:
The investigators will conduct a randomized controlled trial between April 2024 and April 2025 after the ethics committee of the faculty of medicine at Kafr el-Sheik University approves.

The investigators got written informed consent from all eligible patients or their first order of kin before randomization.

The study will be composed of 2 arms atorvastatin arm, which consisted of 300 patients who received 40 mg daily atorvastatin for 3 months, and the rosuvastatin arm consisted of 300 patients who received 20 mg rosuvastatin daily for 3 months, All the patients in the two groups received open-label clopidogrel at a loading dose of 300 mg and then 75 mg daily till the end of the 3 months.

Study Procedures:

Every patient in our study will undergo:

Clinical workup: History, clinical assessment & NIHSS were recorded on admission, day 7, and the Modified Rankin Scale as a follow-up after one week and 3 months.

Detection of Risk Factors & Profiles:

Echocardiography& TOE: in indicated patients ECG Monitoring: daily ECG monitoring will be performed in indicated patients. - Carotid Duplex: carotid duplex in indicated patients.

4- ESR & Lipid Profile& liver functions: All will be tested routinely for all patients.

Imaging Follow-UP Non-contrast CT brain on admission Day 2 MRI: After 2 days of admission, all the patients in this study will have a brain MRI (stroke protocol; T1W, T2W, FLAIR, DWI, T2 Echo Gradient, MRA of all intra-cerebral vessels).

CT brain: Any patient with unexplained clinical deterioration at any time throughout his/her hospital stay will be urgently imaged by CT.

Primary End Point:

The primary efficacy outcome was the rate of new stroke at 90 days

• Secondary End Point: the secondary efficacy outcomes were to evaluate the rates of patients who achieved a significant reduction in NIHSS (decrease of four points or more) at the seventh day or discharge compared to baseline, the rates of a favorable outcome with (mRS = 0-2) after one week and after 90 days in a face-to-face interview in the outpatient clinic, rates of the composite of recurrent stroke, myocardial infarction, and death due to vascular events after 90 days of follow-up, while the secondary safety outcome was the rate of treatment-related acute liver injury assessed by ALT, AST test at 90 days, statin-induced myopathy assessed by CPK at 90 days and other adverse effects assessed by a follow-up questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* males and females aged 18-75
* first-ever moderate and Moderate-to-severe Ischemic Stroke
* Patients are not eligible for rt-PA treatment

Exclusion Criteria:

* The investigators excluded patients who had rapidly resolving symptoms before imaging results, and patients with a known history of persistent or recurrent CNS pathology (e.g., epilepsy, meningioma, multiple sclerosis, history of head trauma with a residual neurological deficit).
* the investigators excluded patients who had clinical seizures at the onset of their stroke, as well as those who had symptoms of any major organ failure, active malignancies, or an acute myocardial infarction within the previous six weeks, and those who were on warfarin, regular ticagrelor during the week before admission, or chemotherapy within the previous year.
* The investigators excluded patients with active peptic ulcers, GIT surgery, bleeding history within the last year, and those with a history of major surgery within the last three months.
* The investigators ruled out of our trial patients who had a known allergy to the study drugs and those with INR > 1.4 or P.T. >18 or blood glucose level < 50 or > 400 mg/DL or blood pressure < 90/60 or > 185/110 mmHg on admission or Platelets < 100,000.
* The investigators excluded pregnant and lactating patients and those with stroke due to venous thrombosis and stroke following cardiac arrest or profuse hypotension ineligible for our trial.
* The investigators excluded patients who were regular users of drugs that affect clopidogrel metabolism, such as ketoconazole, dihydropyridine calcium channel blockers, and rifampin.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2024-04-10 (Actual); Primary Completion 2025-12-10 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
the rate of new stroke at 90 days | 90 days
  Rates of new ischemic stroke occur within three months of treatment. The investigators will perform follow-ups of the patient during visits to the outpatient clinic, and brain CT and/ or MRI will be done if there is suspicion of recurrence of ischemic stroke.

SECONDARY OUTCOMES:
Value of National Institute of Health Stroke Scale (NIHSS) after one week | 7 days
  NIHSS is a tool used by healthcare providers to objectively quantify the impairment caused by a stroke and aid in planning post-acute care disposition.
  It ranges from 0 to 42; the lower the score, the better the stroke condition. The improvement will be counted only if there is a decrease in NIHSS score by four points or more within one week of stroke onset.
value of Modified Rankin Scale (mRS) at one week | 7 days
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability its value ranges from 0 to 6; the lower the score, the better the stroke outcome favorable stroke outcome is considered with mRS value equals two or less.
value of Modified Rankin Scale(mRS) at three months | 3 months
  mRS Measures the degree of disability or dependence in the daily activities of people who have suffered a stroke or other causes of neurological disability its value ranges from 0 to 6; the lower the score, the better the stroke outcome favorable stroke outcome is considered with mRS value equals two or less.
rate of composite recurrent stroke, myocardial infarction, and death due to vascular events | 3 months
  rates of new ischemic stroke, TIA, myocardial infarction, or death from vascular events within three months of treatment the investigators will perform follow-ups of the patient during visits to the outpatient clinic and perform needed investigations such as brain imaging, Electrocardiography, arterial and venous duplex ultrasound imaging.
rate of drug adverse effects | 90 days
  Drug adverse effects: all side effects related to the drugs of our study will be reported
Drug adverse effects: all side effects related to the drugs of our study will be reported | 90 days
  the rate of drug hemorrhagic complications which was evaluated using the PLATO bleeding definition which classified hemorrhagic complications into three types as follows: Major bleeding which had one or more of the following criteria: fatal bleeding, intracranial, intrapericardial, bleeding associated with reduction of hemoglobin > 3-5 g/dl, bleeding required transfusion of two to four units whole blood or PRBCs, bleeding produced hypovolemic shock or severe hypotension that required pressor or surgery; Minor bleeding that required medical intervention to stop or treat bleeding: Minimal bleeding: any bleeding that did not require intervention or treatment such as bruising, bleeding gums, oozing from injection sites.

CONTACTS AND LOCATIONS:
Overall Officials: mohamed G. Zeinhom, MD, Principal Investigator — neurology department kafr el-sheikh university
Locations (1):
- Kafr Elsheikh University Hospital, Kafr ash Shaykh, Egypt

IPD SHARING:
Plan to Share IPD: No
All the data that support the findings of this research will be available from the corresponding author M. Zeinhom upon reasonable request.

REFERENCES:
- [Result] Lopez AD, Mathers CD, Ezzati M, Jamison DT, Murray CJ. Global and regional burden of disease and risk factors, 2001: systematic analysis of population health data. Lancet. 2006 May 27;367(9524):1747-57. doi: 10.1016/S0140-6736(06)68770-9. PMID 16731270
- [Result] Zeinhom MG, Aref HM, El-Khawas H, Roushdy TM, Shokri HM, Elbassiouny A. A pilot study of the ticagrelor role in ischemic stroke secondary prevention. Eur Neurol. 2022;85(1):50-55. doi: 10.1159/000518786. Epub 2021 Aug 30. PMID 34515113
- [Result] Paciaroni M, Ince B, Hu B, Jeng JS, Kutluk K, Liu L, Lou M, Parfenov V, Wong KSL, Zamani B, Paek D, Min Han J, Del Aguila M, Girotra S. Benefits and Risks of Clopidogrel vs. Aspirin Monotherapy after Recent Ischemic Stroke: A Systematic Review and Meta-Analysis. Cardiovasc Ther. 2019 Dec 1;2019:1607181. doi: 10.1155/2019/1607181. eCollection 2019. PMID 31867054